CLINICAL TRIAL: NCT00223444
Title: Clinical-Genetic Variation in GABA/Alcohol Sensitivity
Acronym: GABA-Alcohol
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: John D. Roache/Professor, The University of Texas Health Science Center at San Antonio
Other Study IDs: R21AA013435-03A1 (NIH); AA13435-03A1
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2009-05-01 (Estimated); Status verified 2009-04

CONDITIONS: Alcoholism
Keywords: alcohol; GABA; genetic variation
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specifically, we will determine whether the subject's gene for a brain protein called GABA-alpha-6 is of the "Pro" type or "Ser" type.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Genotype group Pro/Pro
- 2: Genotype group Pro/Ser

SUMMARY:
The purpose of the study is to better understand how genetic factors influence individual sensitivity to alcohol.

DETAILED DESCRIPTION:
We want to find out if there are specific characteristics of a person's genes which will cause them to respond differently to alcohol. Genes are parts of the chromosomes found in the cells of our bodies which control our physical characteristics such the color of our hair, eyes, and other features. Genes are made up of molecules called "DNA" which carry the genetic information we receive from our parents. Just as genes control our physical characteristics, differences in genetic information may also explain why some people are more sensitive to alcohol or have problems drinking too much.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male or female with at least one Hispanic birth parent of Mexican ancestry, 21-25 years of age, and able to read the English-language consent form.
* The subject self-reports current use of 3-30 standard drinks
* The subject is in good physical health as determined by history, physical and laboratory studies of hematology and chemistry
* The subject has a Body Mass Index (BMI) between 20-28
* The subject is not concurrently using psychoactive medication or illicit drugs
* If subject is female, she is not pregnant (determined by weekly urine pregnancy screens), is practicing barrier or chemical methods of birth control, and not nursing babies

Exclusion Criteria:

* The subject meets DSM-IV criteria for any lifetime history of alcohol dependence, or dependence or abuse on any other drug in the past two years excepting tobacco dependence
* The subject currently meets DSM-IV for any other psychiatric (Axis I) disorder, excepting tobacco dependence
* The subject cannot consistently provide alcohol-free breath samples and drug-free urine samples
* The subject uses > 20 cigarettes per day or > 500 mg caffeine per day
* The subject's physical exam, lab tests, and medical histories indicate medical illness requiring treatment or interacting with the alcohol or benzodiazepine treatments
* The subject has a sleep apnea or narrow angle-glaucoma (contraindications for benzodiazepines)
* The subject reports extreme hypersensitivity or allergic reactions to benzodiazepines or unusual hypersensitivity to multiple medications
* The subject is unwilling or unable to consent to all experimental procedures including confidential family history interviews and genetic testing specified by the protocol

Ages: 21 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects who are English-speaking, children of Hispanic ancestry, 21-25 years of age, who drink alcohol but are not alcohol dependent will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2002-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D. Roache, Ph.D., Principal Investigator — The University of Texas Health Science Center at San Antonio